CLINICAL TRIAL: NCT02301403
Title: A Comparative Effectiveness RCT of Optimized Cessation Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Penn State University (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1041 Cessation; A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Smoking Cessation
Keywords: smoking; cessation; tobacco
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices

ARMS (2):
- Modern Usual Care (Active Comparator): Participants assigned to the M-UC will receive 8 weeks of nicotine patch, a single brief, in-person counseling session, a faxed referral to the Wisconsin Tobacco Quit Line (WTQL), and will be signed up for either the QUITNOW app or the Web Coach (both provided by Alere Wellbeing, the vendor that provides the WTQL services).
  Interventions: Drug: Nicotine patch; Behavioral: in-person counseling and quitline counseling
- Abstinence-Optimized Cessation Treatment (Experimental): There are 5 intervention components to include in the AOCT package: 1) Preparation Nicotine Mini-Lozenges; 2) 26-week postquit Combination NRT (nicotine patch + nicotine mini-lozenges); 3) Intensive In-Person Cessation Counseling; 4) Extended Maintenance Counseling Calls; and 5) Automated Adherence Calls.
  Interventions: Drug: Preparation Nicotine Mini-Lozenges; Drug: Combination NRT (nicotine patch + nicotine mini-lozenges); Behavioral: Intensive In-Person Cessation Counseling; Behavioral: Extended Maintenance Counseling Calls; Behavioral: Automated Adherence Calls

INTERVENTIONS:
Drug: Nicotine patch — 8 weeks of nicotine patch
  Arms: Modern Usual Care
Behavioral: in-person counseling and quitline counseling — a single brief, in-person counseling session plus a faxed referral to the Wisconsin Tobacco Quit Line (WTQL), for counseling, including the QUITNOW app and the Website
  Arms: Modern Usual Care
Drug: Preparation Nicotine Mini-Lozenges — Nicotine lozenge prior to attempting to quit smoking
  Arms: Abstinence-Optimized Cessation Treatment
Drug: Combination NRT (nicotine patch + nicotine mini-lozenges) — 26 weeks of combination NRT as part of a quit smoking attempt
  Arms: Abstinence-Optimized Cessation Treatment
Behavioral: Intensive In-Person Cessation Counseling — three 20-min In-person Cessation Counseling sessions
  Arms: Abstinence-Optimized Cessation Treatment
Behavioral: Extended Maintenance Counseling Calls — 8 Maintenance-phase smoking cessation counseling sessions
  Arms: Abstinence-Optimized Cessation Treatment
Behavioral: Automated Adherence Calls — 11 brief, automated calls reminding them to use their medications properly
  Arms: Abstinence-Optimized Cessation Treatment

SUMMARY:
This study is a 2-arm randomized clinical trial (RCT). Participants motivated to quit smoking will be randomized to one of two treatments: 1) a Modern Usual Care (M-UC) vs. 2) Abstinence-Optimized Cessation Treatment (AOCT). The components for the optimized treatment have strong theoretical and empirical support from the investigators previous screening studies.

DETAILED DESCRIPTION:
The ultimate goal of this research is to develop a chronic care treatment package for smokers that will address the challenges and opportunities of each phase of the cessation process - motivation, preparation, cessation, maintenance, and relapse recovery. That is, to develop treatments for smokers not yet ready to quit, those who are preparing to quit, those actively engaged in the quitting process and those who have tried to quit but relapsed. To achieve this goal, this research comprises three distinct research studies, each of which represent a phase in a comprehensive chronic care treatment model for clinical intervention with smokers in the primary care setting: the Motivation Study, the Cessation Study, and the Long-term Quitting Study. The goal of each study is to test and identify effective intervention components for distinct phases of the smoking cessation process. These components will then be combined for future research on the effectiveness of this chronic care treatment package

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years
* smoking >4 cigarettes/day for the previous 6 months
* able to read, write, and speak English
* have reliable phone access and agree to respond to Interactive Voice Response (IVR) phone prompts
* and if currently using NRT, agreeing to use only study medication for the duration of the study
* we will not exclude participants based on their prior use of cessation medication or if they use multiple tobacco products in order to enhance real-world generalization (these will be statistically controlled in analyses)
* not currently attempting to quit smoking
* not intending to quit smoking (defined as no plans to quit in the next month)
* and planning to remain in the intervention catchment area for at least 12 months.

Exclusion Criteria:

* currently taking bupropion or varenicline
* medical contraindications to using NRT including hospitalized (for at least one night) for a stroke, heart attack, congestive heart failure or diabetes in the last 30 days
* diagnosis of or treatment for schizophrenia, a psychotic disorder or bipolar disorder in the last 10 years
* and, if the participant is a woman of childbearing potential, being pregnant or intending to becoming pregnant or unwillingness to use an approved method of birth control during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Piper, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Result] Piper ME, Cook JW, Schlam TR, Jorenby DE, Smith SS, Collins LM, Mermelstein R, Fraser D, Fiore MC, Baker TB. A Randomized Controlled Trial of an Optimized Smoking Treatment Delivered in Primary Care. Ann Behav Med. 2018 Sep 13;52(10):854-864. doi: 10.1093/abm/kax059. PMID 30212849
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- See also: Description: University of Wisconsin Center for Tobacco Research and Intervention — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were patients from seven primary care clinics within two Wisconsin healthcare systems. Smokers who expressed interest in quitting smoking during a clinic visit were referred via the electronic health record (EHR) to the research study. Other smokers from these clinics were recruited via mailings and EHR messaging.
Pre-assignment Details: Primary care patients who passed the phone screen were invited to attend a study visit at their referring clinic to learn more about the study, have eligibility confirmed, and provide written informed consent. No enrolled participants were excluded from the study prior to assignment to groups.
Period: Overall Study
Arm/Group | Modern Usual Care | Abstinence-Optimized Cessation Treatment
Started | 315 | 308
Completed | 287 | 267
Not Completed | 28 | 41
Not completed — Withdrawal by Subject | 28 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modern Usual Care | Abstinence-Optimized Cessation Treatment | Total
Number analyzed (Participants) | 315 | 308 | 623
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.9) | 50.0 (12.5) | 49.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 173 | 357
  Male | 131 | 135 | 266
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 69 | 161
  White | 211 | 220 | 431
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 315 | 308 | 623

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abstinence From Smoking
Description: The outcome measure consists of the number of participants reporting abstinence from smoking at 6 months that is biochemically confirmed (exhaled carbon monoxide < 6 parts per million).
Time Frame: 6 months post treatment
Population: Adult smokers interested in quitting smoking who met inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Modern Usual Care | Abstinence-Optimized Cessation Treatment
Number analyzed (Participants) | 315 | 308
Participants | 19 | 49
Statistical Analysis 1: Comparison: Modern Usual Care; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.69 to 5.14]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for participants using the nicotine patch during 8 weeks of active patch treatment. Adverse event data was collected for participants using the nicotine patch and nicotine mini-lozenge during 26 weeks of active use of these 2 medications post-quit.
Description: Adverse events (AEs) and serious AEs (SAEs) were assessed with the question "Since your last contact with us, have there been any changes in your medical condition or health?"
  * For each nicotine-medication-related symptom reported, severity was assessed and whether the symptom has resolved.
  * For any non-nicotine-medication-related symptoms that are reported as a concern, participants were advised to contact their primary care provider in the clinic as per IRB approval.
Arm/Group | Modern Usual Care | Abstinence-Optimized Cessation Treatment
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/308
Serious Adverse Events (participants affected / at risk) | 0/315 | 0/308
Other Adverse Events (participants affected / at risk) | 66/315 | 139/308
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modern Usual Care (N=315) | Abstinence-Optimized Cessation Treatment (N=308)
Nausea (Gastrointestinal disorders) | 9 (9) | 38 (38)
Headache (Nervous system disorders) | 15 (15) | 15 (15)
Itching or Hives (Immune system disorders) | 22 (22) | 23 (23)
Sore Throat (General disorders) | 1 (1) | 15 (15)
Skin rash (Skin and subcutaneous tissue disorders) | 18 (18) | 33 (33)
Insomnia (Psychiatric disorders) | 7 (7) | 19 (19)
Vivid Dreams (Psychiatric disorders) | 14 (14) | 16 (16)
Hiccups (Gastrointestinal disorders) | 1 (1) | 21 (21)
Mouth Problem (General disorders) | 0 (0) | 15 (15)
Persistent Indigestion (Gastrointestinal disorders) | 7 (7) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT02301403/Prot_SAP_000.pdf
  • Informed Consent Form (2014-12-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT02301403/ICF_001.pdf